CLINICAL TRIAL: NCT05798390
Title: Non-Interventional Study On The Treatment With Bempedoic Acid And/Or Its Fixed-dose Combination With Ezetimibe in Routine Clinical Practice in Patients With Primary Hypercholesterolemia Or Mixed Dyslipidemia
Brief Title: Treatment With Bempedoic Acid And/Or Its Fixed-dose Combination With Ezetimibe in Routine Clinical Practice in Patients With Primary Hypercholesterolemia Or Mixed Dyslipidemia
Acronym: MILOS-Spain
Status: Withdrawn | Type: Observational
Why Stopped: Due to patient availability
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Other Study IDs: DSE-BMP-01-22-EU
Record Dates: First submitted 2023-03-10; First posted 2023-04-04 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Primary Hypercholesterolemia; Mixed Dyslipidemia
Keywords: Primary Hypercholesterolemia; Mixed Dyslipidemia; Bempedoic acid and/or its fixed-dose combination with ezetimibe
MeSH Terms: interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bempedoic acid and/or fixed-dose combination with ezetimibe: Participants with primary hypercholesterolemia or mixed dyslipidemia who received bempedoic acid and/or its fixed-dose combination with ezetimibe.
  Interventions: Drug: Bempedoic acid and/or its fixed dose combination with ezetimibe

INTERVENTIONS:
Drug: Bempedoic acid and/or its fixed dose combination with ezetimibe — This is a non-interventional study. No study medication will be provided as part of this protocol to the patients. Medications will be as prescribed by the treating physician in line with clinical practice.

SUMMARY:
Cardiovascular disease (CVD), especially its management and associated costs, remains a major concern globally. There is a direct correlation between circulating levels of low-density lipoprotein cholesterol (LDL-C) and the incidence of CVD.

This study will assess bempedoic acid/FDC in a real-world clinical setting in adult patients in Spain with hypercholesterolaemia or mixed dyslipidemia.

DETAILED DESCRIPTION:
This non-interventional study will be conducted in order to further understand the potential risks and benefits of bempedoic acid/fixed dose combination (FDC) with ezetimibe in a real-world clinical setting in adult patients with primary hypercholesterolaemia (heterozygous familial and non-familial) or mixed dyslipidaemia and to gain insight into the effectiveness (managing plasma levels of LDL-C) as well as safety (clinical events associated with the treatment modalities). No study medication will be provided as part of this protocol to the patients. Medications will be as prescribed by the treating physician in line with clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate
* At least 18 years of age
* Participants suffering from documented primary hypercholesterolemia or mixed dyslipidemia
* Part 1: For participants treated to a maximum of 6 months or intended to be treated with bempedoic acid/FDC under usual clinical practice conditions and as long as the decision of the physician to start treatment is prior to the inclusion of the participant in the study at the discretion of the physician under no reimbursement conditions at enrollment
* Part 2: For participants treated or intended to be treated with bempedoic acid/FDC under usual clinical practice conditions and as long as the decision of the physician to start treatment is prior to the inclusion of the patient in the study under reimbursed conditions at enrollment
* No contraindications exist according to the SmPC of bempedoic acid/ FDC
* No concurrent participation in an interventional study (Simultaneous participation in other non-interventional studies is possible)
* Life expectancy > 1 -year

Exclusion Criteria:

* As this is a non-interventional study, no explicit exclusion criteria exist in order to avoid selection bias and to allow for documentation of routine clinical practice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of participants treated or intended to be treated with bempedoic acid/ FDC under usual clinical practice conditions and as long as the decision of the physician to start treatment is prior to the inclusion of the patient in the study under no reimbursement conditions (Part 1) or under reimbursed conditions (Part 2) at enrollment and who are unable to reach their LDL-C goals with the maximum tolerated dose of statins or patients who are determined by their treating physician to be statin intolerant.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Summary of Patient Characteristics in Participants With Primary Hypercholesterolaemia or Mixed Dyslipidaemia Following Treatment With Bempedoic Acid And/Or Its Fixed-dose Combination With Ezetimibe | Baseline up to 12 months

SECONDARY OUTCOMES:
Mean Change From Baseline in Systematic Coronary Risk Estimation (SCORE) System Following Treatment With Bempedoic Acid And/Or Its Fixed-dose Combination With Ezetimibe | Baseline up to 12 months
Mean Change From Baseline in Second Manifestations of Arterial Disease (SMART) Score Following Treatment With Bempedoic Acid And/Or Its Fixed-dose Combination With Ezetimibe | Baseline up to 12 months
Mean Change From Baseline in Framingham Risk Score Following Treatment With Bempedoic Acid And/Or Its Fixed-dose Combination With Ezetimibe | Baseline up to 12 months
Mean Change From Baseline in Low-density Lipoprotein Cholesterol Levels | Baseline up to 12 months
Mean Change From Baseline in Atherosclerotic Cardiovascular Disease-Modifying Cholesterol Fragments Levels | Baseline up to 12 months
Mean Change From Baseline in Inflammatory Marker hsCRP Levels | Baseline up to 12 months
Mean Change From Baseline In Uric Acid Levels | Baseline up to 12 months
Number of Participants With Relevant Cardiovascular (CV) Events | Baseline up to 12 months
Number of Participants With Adverse Effects and Adverse Drug Reactions Associated With Bempedoic Acid/FDC Ezetimibe | Baseline up to 12 months
Types of Practitioners Caring for Patients Treated With Bempedoic acid/ FDC with Ezetimibe | Baseline up to 12 months
Number of Participants Who Reported Use of Lipid-modifying Treatments Prior To Or Concomitantly To Receiving Bempedoic Acid/FDC With Ezetimibe | Baseline up to 12 months
Mean Treatment Duration, By Therapy | Baseline up to 12 months
Mean Dosage of Bempedoic Acid/FDC Treatment | Baseline up to 12 months
Mean Length of Prescription Intervals of Bempedoic Acid/FDC Treatment | Baseline up to 12 months
Number of Participants Who Permanently Discontinued or Switched From Bempedoic Acid/FDC Treatment | Baseline up to 12 months
Healthcare Resource Use In Participants Who Were Treated With Bempedoic Acid/FDC With Ezetimibe Treatment | Baseline up to 12 months
Mean Change From Baseline In EuroQol (EQ-5D-5L) and PAM-13 | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo

IPD SHARING:
Plan to Share IPD: No